CLINICAL TRIAL: NCT00004262
Title: PHASE I TRIAL OF GADOLINIUM TEXAPHYRIN (PCI -0120) AS A RADIOSENSITIZER DURING STEREOTACTIC RADIOSURGERY BOOST FOR GLIOBLASTOMA MULTIFORME
Brief Title: Radiation Therapy and Gadolinium Texaphyrin in Treating Patients With Supratentorial Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01400; 99H0239; CDR0000067517; NCI-T99-0041; OSU-9976; OSU-99H0239; U01CA076576 (NIH)
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Surgical Procedures, Operative; Congresses as Topic; Radiotherapy, Conformal; Radiosurgery; motexafin gadolinium; Magnetic Resonance Spectroscopy; Spectrum Analysis

ARMS (1):
- Treatment (motexafin gadolinium, radiotherapy, radiosurgery) (Experimental): Within 5 weeks following surgery, patients receive daily external beam radiotherapy five days a week for 5 weeks. Within 2 weeks following completion of radiotherapy, patients receive gadolinium texaphyrin IV over 2 hours followed 3 hours later by stereotactic radiosurgery. Patients undergoing surgical debulking of tumor prior to external beam radiotherapy receive gadolinium texaphyrin IV over 2 hours, 3 hours prior to surgery in addition to the dose prior to stereotactic radiosurgery.
  Interventions: Procedure: conventional surgery; Radiation: 3-dimensional conformal radiation therapy; Radiation: stereotactic radiosurgery; Drug: motexafin gadolinium; Procedure: magnetic resonance imaging; Procedure: spectroscopy

INTERVENTIONS:
Procedure: conventional surgery
  Other Names: surgery, conventional
Radiation: 3-dimensional conformal radiation therapy
  Other Names: 3D conformal radiation therapy; 3D-CRT
Radiation: stereotactic radiosurgery
Drug: motexafin gadolinium — Given IV
  Other Names: gadolinium texaphyrin; Gd (III) Texaphryin; Gd-Tex; PCI-0120; Xcytrin
Procedure: magnetic resonance imaging — Undergo MRI with both the clinical 1.5 Tesla and research 8 Tesla magnets
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
Procedure: spectroscopy — Undergo plasma-atomic emission spectroscopy (DCP-AES)

SUMMARY:
Phase I trial to study the effectiveness of radiation therapy and gadolinium texaphyrin in treating patients who have supratentorial glioblastoma multiforme. Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as gadolinium texaphyrin may make the tumor cells more sensitive to radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the frequency and grade of toxicity of gadolinium texaphyrin as a radiosensitizer at two dose levels in patients with supratentorial glioblastoma multiforme undergoing stereotactic radiosurgery.

II. Compare the tumor, normal brain, and plasma concentrations of this drug regimen to 1.5 and 8 Tesla MRI images in this patient population.

III. Determine if the 8 Tesla images provide more data than the 1.5 Tesla images in terms of the radiosensitizing drug distribution in the tumor in these patients.

OUTLINE: This is a dose escalation study.

Within 5 weeks following surgery, patients receive daily external beam radiotherapy five days a week for 5 weeks. Within 2 weeks following completion of radiotherapy, patients receive gadolinium texaphyrin IV over 2 hours followed 3 hours later by stereotactic radiosurgery. Patients undergoing surgical debulking of tumor prior to external beam radiotherapy receive gadolinium texaphyrin IV over 2 hours, 3 hours prior to surgery in addition to the dose prior to stereotactic radiosurgery.

Cohorts of 3-6 patients receive escalating doses of gadolinium texaphyrin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

Patients are followed monthly for 3 months, and then every 3 months for 5 years or until death.

PROJECTED ACCRUAL: Approximately 12-18 patients will be accrued for this study within 12-18 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed supratentorial glioblastoma multiforme by stereotactic biopsy, open biopsy, or resection
* Maximum diameter of the tumor mass must be no greater than 4 cm in any dimension, including following debulking surgery
* Tumor must be at least 1.0 cm from the optic chiasm and brainstem
* No oligodendrogliomas, meningiomas, or grade I, II, or III astrocytomas
* No infratentorial tumors
* No multifocal glioblastoma multiforme
* Tumor enhances on MRI
* Must have visible tumor on postoperative MRI following surgical resection
* Performance status - Karnofsky 60-100%
* At least 3 months
* Hemoglobin at least 10.0 g/dL
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 mg/dL
* SGPT no greater than 60 U/L
* Creatinine no greater than 1.3 mg/dL
* Blood urea nitrogen no greater than 24 mg/dL
* Neurological function status 0-3
* No evidence of neuropathy
* No glucose-6-phosphate dehydrogenase deficiency
* No known history of porphyria
* History of prior malignancies allowed
* HIV positive status allowed
* No medical contraindication to MRI imaging (i.e., pacemaker, aneurysm clip, or nonsecure metal fragment close to a critical structure)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during study
* At least 6 weeks since prior chemotherapy
* Concurrent steroids allowed
* No prior radiotherapy to the brain or upper neck
* No greater than 5 weeks since prior surgery and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 1999-11; Primary Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) based on the incidence of dose-limiting toxicity (DLT), as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 2.0 | At the time of stereotactic radiosurgery

SECONDARY OUTCOMES:
Concentration of gadolinium in tumor, normal brain, and plasma by plasma-atomic emission spectroscopy and liquid chromatography with mass spectrometry | At baseline, at 48 hours, and at 2 weeks post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: John Grecula, Principal Investigator — Ohio State University
Locations (1):
- Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio, United States